CLINICAL TRIAL: NCT05112640
Title: Subcuticular Absorbable Staples Versus Conventional Skin Closure in Women Undergoing Cesarean Delivery: A Randomized Control Trial
Brief Title: Subcuticular Absorbable Staples Versus Conventional Skin Closure in Women Undergoing Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Cooper Companies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21-0045
Record Dates: First submitted 2021-10-13; First posted 2021-11-09 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Operative Time; Wound Heal

STUDY DESIGN:
Intervention Model Description: Subjects who agree to participate in the study will be randomized to one of the two groups below in a 1/1 allocation
Who Masked: Outcomes Assessor
Masking Description: Reviewers of wound cosmetics during the post operative time will be blind to the intervention. However, surgeon at the time skin closure and patient will not be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Suture wound closure (Active Comparator): Absorbable sutures for closure of cesarean skin incision using Monocryl manufactured by Ethicon.
  Interventions: Device: Subcuticular monocryl suture manufactured by Ethicon
- Absorbable staple wound closure (Experimental): Staples will be applied as per the manufacturer's instructions intraoperatively using INSORB device manufactured by Cooper Surgical.
  Interventions: Device: INSORB: subcuticular stapling device

INTERVENTIONS:
Device: INSORB: subcuticular stapling device — Under the skin stapling device that delivers absorbable staples
  Arms: Absorbable staple wound closure
Device: Subcuticular monocryl suture manufactured by Ethicon — Under the skin suture placed by hand
  Arms: Suture wound closure

SUMMARY:
Despite the high numbers of cesareans being performed, scientific evidence behind which surgical techniques are best remains uncertain. Our objective is to determine if subcuticular absorbable staples improve operative time and wound cosmetics.

DETAILED DESCRIPTION:
This will be an open-label randomized controlled clinical trial. Women undergoing cesarean delivery will be randomized to have either standard wound closure with Monocryl suture or absorbable subcuticular staples placed by INSORB skin stapling device. The INSORB under the skin stapling device is FDA approved but not currently used as standard of care at UTMB. We will exclude women with intraamniotic infection, immunosuppression, active skin infection, those unlikely to be followed-up after delivery, or unable to provide consent.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Women ≥ 24 weeks viable gestation
* Will be undergoing cesarean delivery

Exclusion Criteria:

* Patient unwilling or unable to provide consent.
* No or very limited prenatal care or a non-resident patient who is unlikely to follow-up after delivery.
* Immunosuppressed subjects: i.e., taking systemic immunosuppressant or steroids (e.g. transplant subjects; not including steroids for lung maturity), HIV with CD4 <200, or other
* Decision not to have skin closure (e.g. secondary wound closure, mesh closure)
* Current skin infection
* Coagulopathy
* High likelihood of additional surgical procedure beyond cesarean (e.g. scheduled hysterectomy, tubal ligation, bowel or adnexal surgery)
* Incarcerated individuals
* Intraamniotic infection
* Subjects participating on other treatment trials or studies that would interfere with the current study's primary outcome.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- John Sealy Hospital at University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to share IPD.

REFERENCES:
- [Background] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Background] Gaertner I, Burkhardt T, Beinder E. Scar appearance of different skin and subcutaneous tissue closure techniques in caesarean section: a randomized study. Eur J Obstet Gynecol Reprod Biol. 2008 May;138(1):29-33. doi: 10.1016/j.ejogrb.2007.07.003. Epub 2007 Sep 6. PMID 17825472
- [Background] Rousseau JA, Girard K, Turcot-Lemay L, Thomas N. A randomized study comparing skin closure in cesarean sections: staples vs subcuticular sutures. Am J Obstet Gynecol. 2009 Mar;200(3):265.e1-4. doi: 10.1016/j.ajog.2009.01.019. PMID 19254586
- [Background] Fick JL, Novo RE, Kirchhof N. Comparison of gross and histologic tissue responses of skin incisions closed by use of absorbable subcuticular staples, cutaneous metal staples, and polyglactin 910 suture in pigs. Am J Vet Res. 2005 Nov;66(11):1975-84. doi: 10.2460/ajvr.2005.66.1975. PMID 16334959
- [Background] Pineros-Fernandez A, Salopek LS, Rodeheaver PF, Drake DB, Edlich RF, Rodeheaver GT. A revolutionary advance in skin closure compared to current methods. J Long Term Eff Med Implants. 2006;16(1):19-27. doi: 10.1615/jlongtermeffmedimplants.v16.i1.30. PMID 16566742
- [Background] Nitsche J, Howell C, Howell T. Skin closure with subcuticular absorbable staples after cesarean section is associated with decreased analgesic use. Arch Gynecol Obstet. 2012 Apr;285(4):979-83. doi: 10.1007/s00404-011-2121-5. Epub 2011 Oct 30. PMID 22037686
- [Background] Schrufer-Poland TL, Ruiz MP, Kassar S, Tomassian C, Algren SD, Yeast JD. Incidence of wound complications in cesarean deliveries following closure with absorbable subcuticular staples versus conventional skin closure techniques. Eur J Obstet Gynecol Reprod Biol. 2016 Nov;206:53-56. doi: 10.1016/j.ejogrb.2016.07.501. Epub 2016 Aug 3. PMID 27632411

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 117 participants signed the consent, 2 participants withdrew. The study terminated early due to the low accrual.
Period: Overall Study
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Started | 59 | 56
Completed | 59 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure | Total
Number analyzed (Participants) | 59 | 56 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5) | 31.1 (5.2) | 30.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 56 | 115
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 40 | 83
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 50 | 48 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 56 | 115

OUTCOME MEASURES:

1. Primary Outcome: Operating Time
Description: Total time for the procedure
Time Frame: Start of surgery through end of skin closure in minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Number analyzed (Participants) | 59 | 56
Minutes | 69.2 (23.7) | 61.9 (21.2)

2. Secondary Outcome: Wound Cosmesis
Description: A digital photograph of the incision will be obtained on wound check visit POD 5-10 days. Each photograph will be evaluated by independent blinded research staff using the Stony Brook Scar Evaluation Scale.These scores are totaled to obtain the final score. The Stony Brook Scar Evaluation will score the scar from 0-5 where 5 shows significant healing.
Time Frame: Time of surgery through six weeks post partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Number analyzed (Participants) | 28 | 22
score on a scale | 3.9 (1.0) | 3.2 (1.2)

3. Secondary Outcome: Number of Participants With Composite Wound Complication
Description: Hematoma, seroma, dehiscence, breakdown of wound, wound infection, endometritis, sepsis, post part fevers
Time Frame: Time of surgery through six weeks post partum
Population: Hematoma, seroma, dehiscence, breakdown of wound, wound infection, endometritis, sepsis, post part fevers
Measure: Count of Participants; unit: Participants
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Number analyzed (Participants) | 59 | 56
Participants | 0 | 2

4. Secondary Outcome: Post Operative Pain
Description: Analog pain scale ranging from 0-10. This is a standard question that nurses as during the post partum period while in the hospital and clinic/nursing visits. The numerical score will be recorded from the patient's chart.
  A score of 0 means no pain, and 10 means the worst pain.
Time Frame: 5-10 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Number analyzed (Participants) | 49 | 52
Units on a scale | .9 (2.2) | .7 (1.9)

5. Secondary Outcome: Number of Adverse Events
Description: Allergic reactions: anaphylaxis, angioedema, skin rashes, including Stevens Johnson and Toxic Epidermal Necrolysis
Time Frame: Time of surgery through six weeks post partum
Measure: Count of Participants; unit: Participants
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Number analyzed (Participants) | 49 | 52
Participants | 0 | 0

6. Secondary Outcome: Use of Resources
Description: Postpartum clinic or emergency room visit within 30 days of delivery, need for imaging or other invasive procedures
Time Frame: Time of surgery through six weeks post partum
Population: Patients who had follow up who were sent to triage for evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Number analyzed (Participants) | 49 | 52
Participants | 0 | 1

7. Secondary Outcome: Skin Closure Time in Minutes
Description: The average of minutes it takes for closure of the skin at time of surgery through weeks post partum.
Time Frame: Time of surgery through six weeks post partum
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
Number analyzed (Participants) | 48 | 43
minutes | 7.6 (2.7) | 4.1 (2.67)

ADVERSE EVENTS:
Time Frame: baseline until the end of the study, up to 6 weeks postpartum
Arm/Group | Suture Wound Closure | Absorbable Staple Wound Closure
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/56
Other Adverse Events (participants affected / at risk) | 0/59 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT05112640/Prot_SAP_000.pdf